CLINICAL TRIAL: NCT05850299
Title: Interest of Performing Two 6-minute Walk Tests at the End of a Pulmonary Rehabilitation Program, in COPD Patients.
Acronym: 2-TM6
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0034 - 2-TM6
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2023-03

CONDITIONS: COPD
Keywords: pulmonary rehabilitation; exercise capacity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In pulmonary rehabilitation, the 6-Minute Walk Test (6MWT) is essential to assess the effects of the program on patients' health. Current guidelines don't recommend to perform two 6MWT at the end of pulmonary rehabilitation. However, a more recent study shows that two 6MWT should be performed at the end of the program to accurately and reliably assess patients' capacities.

The aim of this study is to compare the results of two tests performed at the end of the program by COPD patients to find out whether there is a benefit of performing two 6MWT at the end of pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with stage 2 to 4 (A to D) COPD
* Admitted to pulmonary rehabilitation unit of CH des Pays de Morlaix (CHPM)
* To follow a pulmonary rehabilitation program (4 weeks)
* Patient aged 18 or over
* Patient able to formulate his non-opposition to participate in the study

Exclusion Criteria:

* Contraindication to perform the 6-Minute Walk Test
* Patient under legal protection
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients admitted for pulmonary rehabilitation program in pulmonary rehabilitation unit of CH des Pays de Morlaix (CHPM).
Sampling Method: Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
6 minute walk distance (6MWD) | Two hours
  Comparison of the 6MWD between the first and the second 6-Minute walk test (6MWT) performed at the end of pulmonary rehabilitation program.

CONTACTS AND LOCATIONS:
Overall Officials: Marc BEAUMONT, PhD, Principal Investigator — Centre Hospitalier des Pays de Morlaix
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.